CLINICAL TRIAL: NCT02260388
Title: Patient Assisted Intervention for Neuropathy: Comparison of Treatment in Real Life Situations (PAIN-CONTRoLS)
Brief Title: Patient Assisted Intervention for Neuropathy: Comparison of Treatment in Real Life Situations
Acronym: PAIN-CONTRoLS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001500; PCORI-1306-02496 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Results first posted 2018-07-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-06

CONDITIONS: Cryptogenic Sensory Polyneuropathy
Keywords: CSPN; neuropathy; pain; pain management
MeSH Terms: conditions — Pain; Agnosia | interventions — Nortriptyline; Duloxetine Hydrochloride; Pregabalin; Mexiletine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Nortriptyline (Experimental): Nortriptyline - 25 mg daily for 1 week at bedtime, then 50 mg daily at bedtime for 1 week, then 75 mg daily at bedtime for the remainder of the study.
  Interventions: Drug: Nortriptyline
- Duloxetine (Experimental): Duloxetine - 20 mg daily for 1 week, then 40 mg daily for 1 week, then 60 mg daily for the remainder of the study.
  Interventions: Drug: Duloxetine
- Pregabalin (Experimental): Pregabalin - 100 mg at bedtime for 1 week, then 100 mg 2 times per day for 1 week, then 100 mg 3 times per day for the remainder of the study.
  Interventions: Drug: Pregabalin
- Mexiletine (Experimental): Mexiletine - 200 mg at bedtime for 1 week, then 200 mg 2 times per day for 1 week, then 200 mg 3 times per day for the remainder of the study.
  Interventions: Drug: Mexiletine

INTERVENTIONS:
Drug: Nortriptyline
  Arms: Nortriptyline
Drug: Duloxetine
  Arms: Duloxetine
Drug: Pregabalin
  Arms: Pregabalin
Drug: Mexiletine
  Arms: Mexiletine

SUMMARY:
The purpose of this large comparative effectiveness study led by Richard J. Barohn, MD, of the University of Kansas Medical Center, is to learn about the safety and effectiveness of nortriptyline, duloxetine, pregabalin and mexiletine in treating cryptogenic sensory polyneuropathy (CSPN).

DETAILED DESCRIPTION:
The goal of this research project is to find the best drug for the treatment of pain in patients with CSPN. While the pharmaceutical industry has focused attention on drugs for treating diabetic sensory neuropathy (DSPN), and two drugs are now FDA approved, there have not been any prospective trials in CSPN. And, because there are no studies with CSPN patients, insurance carriers often reject authorizing prescriptions for some drugs for patients with CSPN.

There are four drugs that will be tested in this study: nortriptyline, duloxetine, pregabalin and mexiletine. These drugs are not approved by the FDA for the treatment of CSPN and are considered "investigational" in this study.

There are two periods in this study: Screening/Baseline and Study Drug. During the Screening/Baseline period the researchers will determine eligibility for potential subjects. During the second period, eligible patients who consented to participate will take the study drug. Participants will be randomized to receive one of the four drugs in this study. Participants will know which drug they are taking. Participants will not be allowed to switch groups and receive a different drug during the study.

This study uses an adaptive study design. This means the study can enroll less participants and provide better conclusions. The study design allows the researchers the ability to make changes to the approach of the study or to stop the study early if there are strong results.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cryptogenic sensory polyneuropathy.
* Likert Pain Score of greater than or equal to 4.
* Must not currently be on nortriptyline, duloxetine, pregabalin or mexiletine or similar class of medication for at least 7 days from baseline study visit.

Exclusion Criteria:

* Any medical condition or current medication that would prevent them from taking either nortriptyline, duloxetine, pregabalin or mexiletine.
* Unable to give consent.
* Unable or not willing to comply with the study.
* Other causes for polyneuropathy.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Barohn, MD, Principal Investigator — University of Kansas Medical Center
Locations (46):
- United States (45):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Phoenix Neurological Associates, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado Denver Anschutz Campus, Aurora, Colorado
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - University of Florida - Gainesville, Gainesville, Florida
  - University of Florida Health Science Center - Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Neurological Services of Orlando Research, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - NorthShore Neurological Institute, Glenview, Illinois
  - Indiana University, Indianapolis, Indiana
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Hutchinson Clinic, PA, Hutchinson, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Norton Neurology Services, Louisville, Kentucky
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Spectrum Health System, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Saint Louis University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of Buffalo School of Medicine and Biomedical Sciences, Buffalo, New York
  - Mount Sinai Beth Israel, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Penn State Medical Center, Hershey, Pennsylvania
  - Austin Neuromuscular Center, Austin, Texas
  - Sara Austin, MD, PA, Austin, Texas
  - Seton Brain and Spine Institute, Austin, Texas
  - Texas Neurology, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas
  - University of Texas Health Science Center at Houton, Houston, Texas
  - Grand Medical Clinic, Katy, Texas
  - Neurology Clinic of Central Texas, New Braunfels, Texas
  - University of Texas Health Science Center in San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Barohn RJ, Gajewski B, Pasnoor M, Brown A, Herbelin LL, Kimminau KS, Mudaranthakam DP, Jawdat O, Dimachkie MM; Patient Assisted Intervention for Neuropathy: Comparison of Treatment in Real Life Situations (PAIN-CONTRoLS) Study Team; Iyadurai S, Stino A, Kissel J, Pascuzzi R, Brannagan T, Wicklund M, Ahmed A, Walk D, Smith G, Quan D, Heitzman D, Tobon A, Ladha S, Wolfe G, Pulley M, Hayat G, Li Y, Thaisetthawatkul P, Lewis R, Biliciler S, Sharma K, Salajegheh K, Trivedi J, Mallonee W, Burns T, Jacoby M, Bril V, Vu T, Ramchandren S, Bazant M, Austin S, Karam C, Hussain Y, Kutz C, Twydell P, Scelsa S, Kushlaf H, Wymer J, Hehir M, Kolb N, Ralph J, Barboi A, Verma N, Ahmed M, Memon A, Saperstein D, Lou JS, Swenson A, Cash T. Patient Assisted Intervention for Neuropathy: Comparison of Treatment in Real Life Situations (PAIN-CONTRoLS): Bayesian Adaptive Comparative Effectiveness Randomized Trial. JAMA Neurol. 2021 Jan 1;78(1):68-76. doi: 10.1001/jamaneurol.2020.2590. PMID 32809014
- [Derived] Brown AR, Gajewski BJ, Aaronson LS, Mudaranthakam DP, Hunt SL, Berry SM, Quintana M, Pasnoor M, Dimachkie MM, Jawdat O, Herbelin L, Barohn RJ. A Bayesian comparative effectiveness trial in action: developing a platform for multisite study adaptive randomization. Trials. 2016 Aug 31;17(1):428. doi: 10.1186/s13063-016-1544-5. PMID 27577191

RESULTS

PARTICIPANT FLOW:
Groups:
- Nortriptyline: Nortriptyline - 25 mg daily for 1 week at bedtime, then 50 mg daily at bedtime for 1 week, then 75 mg daily at bedtime for the remainder of the study.
  Nortriptyline
- Duloxetine: Duloxetine - 20 mg daily for 1 week, then 40 mg daily for 1 week, then 60 mg daily for the remainder of the study.
  Duloxetine
- Pregabalin: Pregabalin - 100 mg at bedtime for 1 week, then 100 mg 2 times per day for 1 week, then 100 mg 3 times per day for the remainder of the study.
  Pregabalin
- Mexiletine: Mexiletine - 200 mg at bedtime for 1 week, then 200 mg 2 times per day for 1 week, then 200 mg 3 times per day for the remainder of the study.
  Mexiletine
Period: Overall Study
Arm/Group | Nortriptyline | Duloxetine | Pregabalin | Mexiletine
Started | 134 | 126 | 73 | 69
Completed | 132 | 118 | 70 | 65
Not Completed | 2 | 8 | 3 | 4
Not completed — Lost to Follow-up | 2 | 8 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nortriptyline | Duloxetine | Pregabalin | Mexiletine | Total
Number analyzed (Participants) | 134 | 126 | 73 | 69 | 402
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 91 | 86 | 50 | 41 | 268
  >=65 years | 43 | 40 | 23 | 28 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (12.7) | 59.9 (14.0) | 59.5 (13.6) | 60.7 (13.7) | 60.1 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 68 | 34 | 28 | 189
  Male | 75 | 58 | 39 | 41 | 213
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 4 | 3 | 21
  Not Hispanic or Latino | 126 | 119 | 68 | 66 | 379
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 6 | 4 | 4 | 3 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 11 | 4 | 1 | 26
  White | 113 | 104 | 62 | 64 | 343
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 7 | 3 | 1 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 134 | 126 | 73 | 69 | 402
Patient-Reported Outcomes Measurement Information System (PROMIS) Scale T-Scores [Mean (Standard Deviation); unit: T-Score] — T-score metric: 50 is the mean of a relevant reference population and 10 is the standard deviation (SD). A score of 40 is one SD lower than the mean of the reference population; A score of 60 is one SD higher than the mean of the reference population
  PROMIS Pain Interference Short Form v1.0 8a: Higher scores for pain interference represents worse outcome (more pain interference) PROMIS Fatigue Short Form v1.0 8a Higher scores indicate more fatigue (worse outcome).
  PROMIS Sleep Disturbance Short Form v1.0 8a Higher scores indicate more sleep disturbance (worse outcome).
  T-Score
    PROMIS Pain Interference T-Score | 63.1 (7.0) | 62.4 (6.8) | 63.3 (5.5) | 60.9 (7.9) | 62.5 (6.9)
    PROMIS Fatigue T-Score | 59.6 (3.4) | 59.7 (3.3) | 59.1 (3.7) | 59.7 (3.2) | 59.6 (3.4)
    PROMIS Sleep Disturbance T-Score | 59.1 (9.8) | 60.6 (8.3) | 59.8 (8.7) | 57.0 (11.4) | 59.3 (9.5)
SF12 Health Component Scores [Mean (Standard Deviation); unit: Norm-Based Standardization Score] — SF-12v2® Health Survey Standard The Optum™ SF-12v2® Health Survey is a shorter version of the SF-36v2® Health Survey that uses just 12 questions to measure functional health and well-being from the patient's point of view.
  Survey provides psychometrically-based physical component summary (PCS) and mental component summary (MCS) scores.
  Scores are calibrated so that 50 is the average score or norm, standard deviation = 10.
  Higher scores indicate better health for both mental and physical component summary scores.
  Norm-Based Standardization Score
    Physical Component Score | 38.0 (9.3) | 38.5 (9.3) | 37.9 (9.1) | 41.1 (10.1) | 38.7 (9.4)
    Mental Component Score | 48.0 (10.4) | 46.7 (10.1) | 46.8 (11.3) | 47.2 (11.1) | 47.2 (10.6)
Likert Pain Scale [Mean (Standard Deviation); unit: units on a scale] — Likert Pain Scale - Incremental Scale 0 to 10 with 10 indicating most pain.
  units on a scale | 6.9 (1.5) | 6.7 (1.6) | 6.4 (1.6) | 6.5 (1.7) | 6.7 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Co-Primary Measures: Percent of Patients With at Least a 50% Decrease in Likert Pain Scale From Baseline to Week 12 Follow Up and Percent of Patients That Quit
Description: The final outcome of the study is a combination of two endpoints, efficacy and quit or treatment discontinuation rates. The first endpoint was a patient responder-defined measure of efficacy. A patient was deemed efficacious if a 50% or more reduction was observed in the Likert pain-scale from the baseline visit to the 12 week visit (i.e. 6 at baseline to 3 or less at week 12). The second endpoint was the observed percentage of patients who discontinued treatment prior to the last follow up visit for any reason or were lost to follow up. The utility function, which combines efficacy and quit rates, was used to drive the adaptive randomization, stopping criteria, and final analysis conclusions.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Nortriptyline | Duloxetine | Pregabalin | Mexiletine
Number analyzed (Participants) | 134 | 126 | 73 | 69
Participants
  Efficacious and Non-Quit | 34 | 29 | 11 | 14
  Non-Efficacious and Non-Quit | 49 | 50 | 31 | 15
  Quit | 51 | 47 | 31 | 40

2. Secondary Outcome: SF12 Health Composite Scores
Description: SF-12v2® Health Survey Standard The Optum™ SF-12v2® Health Survey is a shorter version of the SF-36v2® Health Survey that uses just 12 questions to measure functional health and well-being from the patient's point of view.
  Survey provides psychometrically-based physical component summary (PCS) and mental component summary (MCS) scores.
  Scores are calibrated so that 50 is the average score or norm, standard deviation = 10.
  Higher scores indicate better health for both mental and physical component summary scores.
Time Frame: 12 weeks
Population: No secondary data were collected for participants who 'Quit' taking the study medication prior to study completion. Thus, only participants that were deemed efficacious and non-quit, or non-efficacious and non-quit at the primary outcome were collected and analyzed for the secondary outcome measure.
Measure: Mean (Standard Deviation); unit: Norm-Based Standardization Score
Arm/Group | Nortriptyline | Duloxetine | Pregabalin | Mexiletine
Number analyzed (Participants) | 83 | 79 | 42 | 29
Norm-Based Standardization Score
  Mental Component Score | 51.0 (8.9) | 50.9 (9.9) | 47.2 (11.2) | 51.3 (10.8)
  Physical Component Score | 42.8 (8.7) | 42.1 (9.5) | 40.0 (8.2) | 43.7 (9.6)

3. Secondary Outcome: PROMIS Pain Interference Short Form v1.0 8a T Score
Description: Higher scores for pain interference represents worse outcome (more pain interference) T-score metric: 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
  On the T-score metric: A score of 40 is one SD lower than the mean of the reference population; A score of 60 is one SD higher than the mean of the reference population.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Nortriptyline | Duloxetine | Pregabalin | Mexiletine
Number analyzed (Participants) | 83 | 79 | 42 | 29
T-Score | 56.4 (8.4) | 56.5 (8.3) | 60.0 (7.5) | 54.5 (8.8)

4. Secondary Outcome: PROMIS Fatigue Short Form v1.0 8a
Description: Higher scores for fatigue represents worse outcome (more fatigue). T-score metric: 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
  On the T-score metric: A score of 40 is one SD lower than the mean of the reference population; A score of 60 is one SD higher than the mean of the reference population.
Time Frame: 12 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Nortriptyline | Duloxetine | Pregabalin | Mexiletine
Number analyzed (Participants) | 83 | 79 | 42 | 29
T-Score | 53.6 (9.5) | 55.4 (10.2) | 56.7 (10.6) | 51.6 (10.7)

5. Secondary Outcome: PROMIS Sleep Disturbance Short Form v1.0 8a
Description: Higher scores for sleep disturbance represents worse outcome (more sleep disturbance).
  T-score metric: 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
  On the T-score metric: A score of 40 is one SD lower than the mean of the reference population; A score of 60 is one SD higher than the mean of the reference population.
  Higher scores equals more of the concept being measured
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Nortriptyline | Duloxetine | Pregabalin | Mexiletine
Number analyzed (Participants) | 83 | 79 | 42 | 29
T-Score | 58.9 (2.5) | 58.9 (2.6) | 58.3 (2.3) | 59.1 (2.0)

ADVERSE EVENTS:
Time Frame: 12 Weeks Post Randomization
Arm/Group | Nortriptyline | Duloxetine | Pregabalin | Mexiletine
All-Cause Mortality (participants affected / at risk) | 0/134 | 0/126 | 0/73 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/134 | 0/126 | 0/73 | 0/69
Other Adverse Events (participants affected / at risk) | 75/134 | 59/126 | 29/73 | 27/69
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nortriptyline (N=134) | Duloxetine (N=126) | Pregabalin (N=73) | Mexiletine (N=69)
Dry Mouth (Nervous system disorders) | 27 | 3 | 1 | 3
Drowsiness/Sleepiness (Nervous system disorders) | 16 | 7 | 8 | 3
Nausea (Ear and labyrinth disorders) | 3 | 11 | 1 | 6
Insomnia (General disorders) | 5 | 12 | 1 | 2
Fatigue (Nervous system disorders) | 7 | 8 | 3 | 1
Bloating/Constipation (Gastrointestinal disorders) | 10 | 3 | 1 | 2
Headache (Nervous system disorders) | 4 | 2 | 2 | 1
Other (Nervous system disorders) | 3 | 13 | 12 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT02260388/Prot_SAP_000.pdf